CLINICAL TRIAL: NCT00538395
Title: Intensive Sequential Chemotherapy With Adriamycin Taxol and Cytoxan in the Treatment of Locally Advanced Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAC #981-020
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Paclitaxel; Cyclophosphamide

INTERVENTIONS:
Drug: Adriamycin, Taxol and Cytoxan — Chemotherapy

SUMMARY:
Intensive sequential chemotherapy with Adriamycin Taxol and Cytoxan in the treatment of locally advanced breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced breast cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-09; Primary Completion 2012-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Effectiveness | overall

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Ezzat, MD, Principal Investigator — KFSH&RC, Riyadh, Saudi Arabia